CLINICAL TRIAL: NCT05685927
Title: Understanding Muscular Deficits of Diabetic Myopathy
Brief Title: Investigating Muscle Failure in Diabetic Myopathy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DM2021AS
Record Dates: First submitted 2023-01-03; First posted 2023-01-17 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Obesity; Chronic Hyperglycaemia; Weight Loss; Diabetic Myopathy; Sarcopenia
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Weight Loss; Sarcopenia | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Non-obese participants with dysregulated type 1 diabetes
  Interventions: Drug: 6-months of medically assisted glycemic improvement
- Non-obese participants with dysregulated type 2 diabetes
  Interventions: Drug: 6-months of medically assisted glycemic improvement
- Obese participants with type 2 diabetes
  Interventions: Procedure: Bariatric surgery
- Obese participants without type 2 diabetes
  Interventions: Procedure: Bariatric surgery
- Healthy control participants

INTERVENTIONS:
Drug: 6-months of medically assisted glycemic improvement — Administrated by the clinic at Steno Diabetes Center, Aarhus, Denmark
  Groups: Non-obese participants with dysregulated type 1 diabetes; Non-obese participants with dysregulated type 2 diabetes
Procedure: Bariatric surgery — Participants are examined prior to and 1 year following bariatric surgery in the Central Region, Denmark
  Groups: Obese participants with type 2 diabetes; Obese participants without type 2 diabetes

SUMMARY:
The goal of this observational study is to assess if diabetes and obesity are independently related to functional and structural muscle deficits, and how muscular deficits relate to metabolic properties of diabetes and obesity. All studies will include clinical muscle strength and contractile examinations, functional tests, and MR imaging and spectroscopy techniques.

The main questions this project aims to answer are:

1. Is chronic hyperglycemia in type 1 and 2 diabetes associated with functional and structural deficits of skeletal muscles unrelated to the presence of neuropathy?
2. Is obesity associated with functional and structural impairments of skeletal muscles unrelated to the presence of type 2 diabetes ?
3. Does weight loss improve muscle metabolic flexibility and economy and modify skeletal muscle function and structure in obese subjects with and without type 2 diabetes?

The project will include three studies, intended to answer the hypotheses listed above:

Study 1: Evaluation of functional and structural muscular deficits of diabetic myopathy in relation to prolonged hyperglycemia prior to and 6 months following glycemic improvement in patients with type 1 and 2 diabetes

Study 2: Functional and structural muscular deficits in severely obese subjects with and without type 2 diabetes prior to assisted weight loss.

Study 3: Changes in functional and structural muscle properties following assisted weight loss in severely obese subjects with and without type 2 diabetes - a 1-year follow-up study.

ELIGIBILITY:
Inclusion Criteria:

Study 1:

* Age: 18-60 years
* BMI: 18.5 - 39, minimum weight = 50kg
* Chronic hyperglycemia: HbA1c of ≥ 70 mmol/mol with a duration of ≥ 2 months prior to enrollment
* Physical activity: Less than 3 x 60 min of structured physical activity per week

Study 2 & 3:

* Age: 25-60 years
* BMI: ≥ 35
* Physical activity: Less than 3 x 60 min of structured physical activity per week

Healthy Control Participants:

* Age: 18-60 years
* BMI: 18.5 - 30, minimum weight = 50kg
* Physical activity: Less than 3 x 60 min of structured physical activity per week

Exclusion Criteria:

Study 1, 2, 3 and healthy controls:

* Diabetic neuropathy with expected motor deficits
* Uncontrolled cardiovascular or pulmonary disease, peripheral vascular disease, osteoarthropathy of the lower extremity, or any neurological og rheumatological disease which may affect muscle function, as well as any other disease that may effect ones ability to perform physical activity.
* Any Magnetic Resonance contraindications
* Any condition that by the principal investigator is expected to affect the participants ability to execute the study elements

Specifically for healthy control participants:

* The presence of diabetes or pre-diabetes (HbA1c ≥42 mmol/mol)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consist of participants with type 1 diabetes (study 1) and participants with obesity and/or type 2 diabetes (study 1 and 2). Participants will be included at the Dept. of Endocrinology and Steno Diabetes Center Aarhus, Aarhus University Hospital, Denmark. Healthy control participants will be recruited by advertising in local media and at dedicated participant recruitment homepages.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Baseline: Evaluating the presence of sarcopenia in relation to the presence of hyperglycemia and/or obesity | The prevalence of sarcopenia in participants with diabetes and hyperglycemia (study 1) or obesity (study 2) as compared to healthy control participants at baseline
  The presence of sarcopenia is assessed based on recommended methods including measures of muscle strength (Biodex Dynamometer), muscle quantity and quality (MRI), and physical performance tests.
Baseline: Skeletal muscle Force-velocity assessment in relation to the presence of hyperglycemia and/or obesity | The force-velocity relationship in participants with diabetes and hyperglycemia (study 1) or obesity (study 2) as compared to healthy control participants at baseline
  Assessed by isokinetic knee-extension and dorsal flexion on a Biodex Dynamometer at increasing angular-velocities
Baseline: Assessment of skeletal muscle fatigue in relation to the presence of hyperglycemia and/or obesity | Fatigue in participants with diabetes and hyperglycemia (study 1) or obesity (study 2) as compared to healthy control participants at baseline
  Assessed by a fatiguing isotonic protocol for knee-extension and dorsal flexion on a Biodex Dynamometer including twitch-parameters of knee-extensors
Changes in skeletal muscle force-velocity relationship with weight-loss or glycemic improvement | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3
Changes in skeletal muscle fatigue in relation to weight-loss or glycemic improvement | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3
Changes in parameters defining sarcopenia in relation to weight-loss or glycemic improvement | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3

SECONDARY OUTCOMES:
31P MRS: Skeletal muscle bioenergetics and metabolic economy | Bioenergetics and metabolic economy in participants with diabetes and hyperglycemia (study 1) or obesity (study 2) as compared to healthy control participants at baseline
  Assessed by phosphorus magnetic resonance spectroscopy (31P MRS) performed during an isotonic fatiguing exercise in a 3T MR-scanner
31P MRS: Changes of skeletal muscle bioenergetics and metabolic economy in relation to weight-loss or glycemic improvement | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3
  Assessed by phosphorus magnetic resonance spectroscopy (31P MRS) performed during an isotonic fatiguing exercise in a 3T MR-scanner
ENG assessment of neuropathic changes | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3
  ENG is assessed in the Sural, Tibial and Peroneal nerve
Correlation analyses of primary measures with metabolic parameters including insulin resistance, HbA1c, metabolic economy, bioenergetics, and low-grade systemic inflammation (hs-CRP) | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3

OTHER OUTCOMES:
EMG assessment of myopathic changes | Change from baseline to follow-up at an average of 6 months for study 1 and 12 months for study 3
  Will be assessed in knee extensors and/or dorsal flexors on a subgroup of participants demonstrating significant fatigue during primary measures

CONTACTS AND LOCATIONS:
Overall Officials: Anders Stouge, MD, PhD-student, Principal Investigator — Aarhus University, Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Denmark, Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlies results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code